CLINICAL TRIAL: NCT05044429
Title: Postoperative Pain Control With Systemic Lidocaine vs. Regional Anesthesia in Renal Transplant Patients
Brief Title: Postoperative Pain Control Following Renal Transplant
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of interest for continuing on by PI and issues with IRB
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Eric Heinz, Associate Professor of Anesthesiology and Critical Care, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCR202221
Record Dates: First submitted 2021-04-13; First posted 2021-09-14 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Kidney Transplant; Complications; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Intravenous Lidocaine (Experimental)
  Interventions: Drug: Intravenous Lidocaine
- Transversus abdominis plane (TAP) block (Active Comparator)
  Interventions: Drug: Transversus abdominis plane (TAP) block
- Quadratus Lumborum (QL) Block (Active Comparator)
  Interventions: Drug: Quadratus Lumborum (QL) Block

INTERVENTIONS:
Drug: Intravenous Lidocaine — Patient will receive intravenous lidocaine 1.0-1.5 mg/kg/hour for 48 hours post-operatively in addition to standard of care (patient-controlled analgesia (PCA) pump)
  Arms: Intravenous Lidocaine
Drug: Transversus abdominis plane (TAP) block — Subject will receive 0.2% Ropivacaine at 6-10ml/hour through transversus abdominis plane (TAP) block for up to five days post-operatively in addition to standard of care (patient-controlled analgesia (PCA) pump)
  Arms: Transversus abdominis plane (TAP) block
Drug: Quadratus Lumborum (QL) Block — Subject will receive 0.2% Ropivacaine at 6-10ml/hour through quadratus lumborum (QL) block for up to five days post-operatively in addition to standard of care (patient-controlled analgesia (PCA) pump)
  Arms: Quadratus Lumborum (QL) Block

SUMMARY:
This study aims to compare the effectiveness of a regional anesthetic block vs systemic intravenous (IV) lidocaine in controlling post-operative pain in kidney transplantation patients. Regional anesthetic blocks and lidocaine infusions are effective alternatives to opioid medications and are already in use at many institutions. However, there has been no prospective study comparing their effectiveness when used in conjunction with the current standard of care patient controlled analgesia (PCA) pumps. This study is a prospective, randomized evaluation of both treatment methods.

DETAILED DESCRIPTION:
Adequate postoperative pain control is an important part of the patients' recovery. Renal transplant patients often have multiple comorbidities, that when combined with poorly controlled postoperative pain, can lead to tachycardia, hypertension, and increased risk of respiratory complications, which can in turn affect overall recovery and graft survival.

The use of patient-controlled analgesia (PCA) pumps is currently considered the standard of care in treating surgical pain in the immediate postoperative period. Although a traditional mainstay of therapy, opioids have an unfavorable side effect profile that includes respiratory depression, nausea, postoperative ileus, sedation, and pruritus. Additionally, long-term opioid use is linked with opioid tolerance, addiction, and patient death. Patients that have high-level opioid use in the first year posttransplant have been found to have high rates of death and all-cause graft failure.

Recently, there has been a shift in post-operative pain management to utilize a multimodal approach of both non-pharmacologic and pharmacologic therapies. As a result, the use of other non-opioid therapies, such as lidocaine infusions and regional anesthetic techniques, like transverse abdominis plane blocks, have recently increased in popularity in perioperative pain management of renal transplant patients.

Intravenous lidocaine has an off label indication as analgesic and has good evidence for use in other areas such as colorectal surgery, trauma and orthopedics. Lidocaine infusions have a strong record of safety with relatively benign adverse side effects. Although data is promising, there is little established evidence of perioperative lidocaine infusions in renal transplant populations.

Transverse abdominis plane (TAP) blocks and quadratus lumborum (QL) blocks have emerged as a significant regional technique in the application of multimodal analgesia for abdominal surgeries. Historically, TAP and QL catheters are avoided due to concern about infection near the operative site in immunosuppressed transplant patients. Establishing intravenous lidocaine as an effective treatment option will allow physicians to avoid the side effects of opioids and the infection risks of TAP and QL catheter blocks.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral renal transplant

Exclusion Criteria:

* History of chronic pain, chronic opioid use, or opioid use disorder
* Cardiac arrythmia, cardiac failure
* Hepatic Failure
* Local anesthetic allergy (allergy to lidocaine and ropivacaine)
* Complicated surgical course including intraoperative damage to other organs (bowel)
* Return to operating room within 72hours

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farag E, Guirguis MN, Helou M, Dalton JE, Ngo F, Ghobrial M, O'Hara J, Seif J, Krishnamurthi V, Goldfarb D. Continuous transversus abdominis plane block catheter analgesia for postoperative pain control in renal transplant. J Anesth. 2015 Feb;29(1):4-8. doi: 10.1007/s00540-014-1855-1. Epub 2014 Jun 5. PMID 24898186
- [Background] Beaussier M, Delbos A, Maurice-Szamburski A, Ecoffey C, Mercadal L. Perioperative Use of Intravenous Lidocaine. Drugs. 2018 Aug;78(12):1229-1246. doi: 10.1007/s40265-018-0955-x. PMID 30117019
- [Background] Rahendra R, Pryambodho P, Aditianingsih D, Sukmono RB, Tantri A, Melati AC. Comparison of IL-6 and CRP Concentration Between Quadratus Lumborum and Epidural Blockade Among Living Kidney Donors: A Randomized Controlled Trial. Anesth Pain Med. 2019 Apr 28;9(2):e91527. doi: 10.5812/aapm.91527. eCollection 2019 Apr. PMID 31341831

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Started | 19 | 7 | 5
Completed | 19 | 7 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block | Total
Number analyzed (Participants) | 19 | 7 | 5 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 6 | 5 | 29
  >=65 years | 1 | 1 | 0 | 2
Age, Continuous [Mean (Full Range); unit: years] | 49.1 [25 to 69] | 49.8 [24 to 76] | 52.2 [32 to 64] | 49.8 [24 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 1 | 15
  Male | 9 | 3 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 0 | 5
  Not Hispanic or Latino | 16 | 4 | 5 | 25
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 3 | 5 | 24
  White | 0 | 2 | 0 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants] — Population: trial was terminated before analysis of data

OUTCOME MEASURES:

1. Primary Outcome: Opioid Utilization (12 Hour Post-operative)
Description: We are measuring oral morphine equivalents to assess for study intervention efficacy at 12 hours after surgery
Time Frame: 12 hours after surgery
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Opioid Utilization (24 Hour Post-operative)
Description: We are measuring oral morphine equivalents to assess for study intervention efficacy at 24 hours after surgery
Time Frame: 24 hours after surgery
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Opioid Utilization (36 Hour Post-operative)
Description: We are measuring oral morphine equivalents to assess for study intervention efficacy at 36 hours after surgery
Time Frame: 36 hours after surgery
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Opioid Utilization (48 Hour Post-operative)
Description: We are measuring oral morphine equivalents to assess for study intervention efficacy at 48 hours after surgery
Time Frame: 48 hours after surgery
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

5. Primary Outcome: Pain Level (12 Hour Post-operative)
Description: Measured using visual analog scale (0-10), 0 is the best and 10 is the worst score at 12 hours after surgery
Time Frame: 12 hours after surgery
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

6. Primary Outcome: Pain Level (24 Hour Post-operative)
Description: Measured using visual analog scale (0-10), 0 is the best and 10 is the worst score at 24 hours after surgery
Time Frame: 24 hours after surgery
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

7. Primary Outcome: Pain Level (36 Hour Post-operative)
Description: Measured using visual analog scale (0-10), 0 is the best and 10 is the worst score at 36 hours after surgery
Time Frame: 36 hours after surgery
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

8. Primary Outcome: Pain Level (48 Hour Post-operative)
Description: Measured using visual analog scale (0-10), 0 is the best and 10 is the worst score at 48 hours after surgery
Time Frame: 48 hours after surgery
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Subjects With Postoperative Sepsis
Description: We will be assessing for a number of patients with post-operative infection that requires intravenous antibiotics
Time Frame: Through hospital discharge, approximately three days
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Number of Acute Rejection of Renal Transplant
Description: Occurs when the immune system identifies a grafted organ as foreign and attacks it
Time Frame: Up to one week
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Number of Subjects With Local Anesthetic Systemic Toxicity (LAST)
Description: A life-threatening adverse reaction resulting from local anesthetic reaching significant systemic circulating levels
Time Frame: Through hospital discharge, approximately four days
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Number of Patients Who Need Continuous Veno-venous Hemodiafiltration (CVVHDF) After Renal Transplant
Description: Temporary treatment for patients with acute renal failure
Time Frame: By time of hospital discharge, approximately four days
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Number of Patients With Symptoms of Opioid Toxicity After Renal Transplant
Description: Opioid toxicity requiring naloxone
Time Frame: Through hospital discharge, approximately four days
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Number of Patients With Ileus After Renal Transplant
Description: Painful obstruction of the ileum or other part of the intestine
Time Frame: Through hospital discharge, approximately four days
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Total Length of Hospital Stay
Description: Transplant time to discharge time
Time Frame: Through hospital discharge, approximately four days
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Length of Intensive Care Unit Stay
Description: Number of days spent in the intensive care unit following transplant
Time Frame: Through hospital discharge, approximately four days
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Vital Status
Description: Alive or dead at time of hospital discharge
Time Frame: Through hospital discharge, approximately four days
Population: trial was terminated before the outcome measure data were collected
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 7.5 months
Arm/Group | Intravenous Lidocaine | Transversus Abdominis Plane (TAP) Block | Quadratus Lumborum (QL) Block
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/19 | 0/7 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT05044429/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT05044429/ICF_001.pdf